CLINICAL TRIAL: NCT00101569
Title: Aripiprazole Oral Acceptability Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN138-091
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2008-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: Aripiprazole
- A2 (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 15 -30 mg, once daily, 2 weeks (days 1 -14).
  Other Names: Abilify
  Arms: A1
Drug: Aripiprazole — Oral Solution, Oral, 15-30 ml, once daily, 1 week (days 15 -21).
  Other Names: Abilify
  Arms: A2

SUMMARY:
The purpose of this trial is to study liquid aripiprazole in patients with stable schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients currently receiving aripiprazole or other antipsychotic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59
Dates: Start 2004-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - Local Institution, Anaheim, California
  - Local Institution, National City, California
  - Local Institution, North Miami Beach, Florida
  - Local Institution, Overland Park, Kansas
  - Local Institution, Staten Island, New York
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Falls Church, Virginia